CLINICAL TRIAL: NCT04190329
Title: Feasibility of an Extended Test Battery and Influencing Factors for Detecting Frailty
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: Frailty-Testing
Record Dates: First submitted 2019-11-28; First posted 2019-12-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 10 non-frail (robust) study patients: Patients fulfill 0 criteria according to modified Fried frailty score.
- 10 pre-frail study patients: Patients fulfill 1-2 criteria criteria according to modified Fried frailty score.
- 10 frail study patients: Patients fulfill 3, 4 or 5 criteria according to modified Fried frailty score.

SUMMARY:
The aim of the prospective study is to assess the feasibility of a screening and baseline measurement protocol that is planned for a main study (PRÄP-GO) in a collective of 30 patients ageing 70+ scheduled for elective surgery. Comprehensive geriatric assessment scores and modified Fried frailty phenotype component evaluation are performed in all patients at baseline before elective surgery. The assessment of cognitive tests is conducted with a battery of neuropsychological tests, computer-based tests from the Cambridge Neuropsychological Test Automated Battery [CANTAB®] and non-computer based tests. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) represent robust (0), pre-frail (1-2), and frail (3-5) health status. 10 patients without Frailty, 10 patients with Pre-Frailty and 10 patients with Frailty should be analyzed in this study and receive further comprehensive geriatric assessment testing up to seven days after surgery/discharge (before 7 postoperative days).

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 70 years
* Male and female patients
* Patient eligible for inclusion: by the patient, preoperatively
* elective surgery
* Expected anesthesia duration> 60min

Exclusion criteria:

* Severe cardiological or pulmonary disease (NYHA IV, Gold IV)
* Intracranial interventions
* Moribund patients (palliative situation)
* Not enough language skills
* Non-consenting patients
* Participation in another prospective intervention study for study inclusion or throughout the study period.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing elective surgery aged ≥70 years, including 10 patients without Frailty, 10 patients with Pre-Frailty and 10 patients with Frailty.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Duration to run the test battery | 1 day (Once only at screening)
  The duration of the screening test battery is measured with a stopwatch.

SECONDARY OUTCOMES:
Acceptance of test battery | 1 day (Once only at screening)
  The study patient´s acceptance of the screening test battery is measured with a questionnaire.
Problems to conduct the test battery | 1 day (Once only at screening)
  Problems while performing the test battery are categorized according to a standardized protocol.
Change in pain | Baseline, day 3 after surgery and discharge or day 7 after surgery
  Pain is measured with a pain score, a higher score indicates more pain.
Intelligibility of the patient Diary 1 | Up to day 7 after surgery
  Number of completed items
Intelligibility of the patient Diary 2 | Up to day 7 after surgery
  Number of completed days
Intelligibility of the patient Diary 3 | Up to day 7 after surgery
  Coherence of the diary with clinical patient record
Implementation rate of the patient Diary 3 | Up to day 7 after surgery
Handgrip strength | Baseline, day 3 after surgery and discharge or day 7 after surgery
  Handgrip strength measured using a Dynamometer.
Mobility | Baseline, day 3 after the operation and discharge or day 7 after surgery
  Mobility is measured using the Charité Mobilitäts-Index (CHARMI®).
Nutritional status 1 | Baseline and discharge or day 7 after surgery
  Nutritional status 1 is measured using serum albumin.
Nutritional status 2 | Baseline and discharge or day 7 after surgery
  Nutritional status 2 is measured using arm circumference.
Nutritional status 3 | Baseline and discharge or day 7 after surgery
  Nutritional status 3 is measured using calf circumference.
Nutritional status 4 | Baseline and discharge or day 7 after surgery
  Nutritional status 4 is measured using the Mini Nutritional Assessment - Short Form (MNA®-SF).
Intra- and postoperative organ complications | Up to 7 days after surgery
Length of intensive care unit stay | Participants will be followed for the duration of hospital stay, an expected average of 1 day.
Length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days.

OTHER OUTCOMES:
Cognitive Status | 1 day (Once only at screening)
  Neuropsychological testing
Depression | 1 day (Once only at screening)
  The assessment of Depression is measured with the - Patient Health Questionnaire (PHQ-8)
Frailty | 1 day (Once only at screening)
  Frailty is operationalized using modified Fried frailty criteria. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) represent robust (0), pre-frail (1-2), and frail (3-5) health status.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité Univerisitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No